CLINICAL TRIAL: NCT05704335
Title: INFLUENCEF STUDY: Epidemiology, Risk Factors and Clinical Phenotype of Headache Associated With Influenza Infection
Brief Title: InfluenCEF Study: Study on the Headache Associated With Influenza Infection
Acronym: INFLUENCEF
Status: Recruiting | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Collaborators: Red Centinela Sanitaria de Castilla y León (RCSCYL) (Unknown); Centro Nacional de Gripe de Valladolid (CNGV) (Unknown); Dirección General de Salud Pública de la Consejería de Sanidad de la Junta de Castilla y León (Unknown)
Responsible Party: Principal Investigator, David García Azorín, David García-Azorín, MD, PhD, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI 22- 2884
Record Dates: First submitted 2022-12-23; First posted 2023-01-30 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Headache Disorders; Influenza -Like Illness; Head Pain; Migraine; Viral Infection
Keywords: Headache disorders; Secondary headache; Virus diseases; Epidemiology; Influenza
MeSH Terms: conditions — Headache Disorders; Headache; Migraine Disorders; Virus Diseases; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab with sterile swab samples are sent to local laboratories where molecular analysis is performed by PCR to detect influenza viruses and other respiratory pathogens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with headache during the course of influenza: Patients with influenza infection who experience new-onset headache during the course of the disease, or a two-fold worsening of a prior headache disorder, according to the International Classification of Headache Disorders
  Interventions: Other: Questionnaire administration

INTERVENTIONS:
Other: Questionnaire administration — A trained physician will administer a structured questionnaire

SUMMARY:
The goal of this observational analytic study with a cohort desing is to evaluate the epidemiology, risk factors and clinical phenotype of headache during Influenza infection. The study will be done in collaboration with the Healthcare Sentinel Network of Castile and Leon (Red Centinela Sanitaria de Castilla y León, RCSCYL) and the National Influenza Center of Valladolid (CNGV). First, the historical data of the VIGIRA network of the 2010-2022 flu seasons will be analyzed, assessing the epidemiology and risk factors of headache during Influenza infection; and second, a study with a case series design with prospective follow-up will be carried out for the incident cases of the 2022-2023 and 2023-2024 Influenza seasons, evaluating the clinical phenotype and the duration of the headache.

DETAILED DESCRIPTION:
Respiratory tract infections are the second global cause of disability-adjusted life years and represent a higher cost than illnesses such as heart failure, asthma, or migraine. The influenza virus is responsible for 11.5% of episodes of lower respiratory tract infections, causing 650,000 deaths per year. In Spain, in the period prior to COVID-19, the incidence rate of influenza infection was estimated in 2,069 cases per 100,000 inhabitants and year. Between 2001 and 2018, the seasonal transmissibility of influenza viruses has varied depending on diverse factors, such as the type/subtype of influenza, the dominant or codominance of multiple strains, and the timing of the epidemic. The diagnosis of the infection has evolved in the latest years, allowing to monitor the epidemics and elaborate sanitary programs that permit its control and management.

The Healthcare Sentinel Network of Castile and Leon - Red Centinela Sanitaria de Castilla y León (RCSCYL) carries out active influenza surveillance since the 1996-1997 season, and additionally, since the 2020 monitors other Acute Respiratory Infections (ARI) (VIGIRA system) in collaboration with the National Influenza Center of Valladolid (CNGV), the department of Microbiology of the University Clinical Hospital of Valladolid. This program works in collaboration with the National Influenza Surveillance System of Spain (SVGE), integrated into the European Influenza Surveillance Network (EISN). Active monitoring is done by 100 healthcare providers covering a 60,000 population.

The current VIGIRA program includes those patients who belong to a quota of a sentinel general practitioner or pediatrician that are evaluated in primary care (PC) setting due to an ARI. The World Health Organization (WHO) definition of ARI, as acute onset of at least one of the following four respiratory symptoms: cough, sore throat, shortness of breath, coryza, and a clinician's judgement that the illness is due to an infection. The definition states that ARIs may present with or without fever. During the 2021-2022 season, until June 12, 2022, the rate of ARIs has been of 43,841 cases per 100,000 population.

Influenza is defined as the clinical syndrome caused by influenza family viruses' infection. It is characterized by a combination of respiratory and systemic symptoms. Headache is one of the most frequent systemic symptoms, although the number of specific studies is very scarce. Up to now, only two studies that included 37 and 279 patients have shown prevalence rates for this symptom between 32.4% and 60%.

In 2008, the criteria that defines the influenza-like illness was modified, to an acute respiratory illness with onset during the last 7 days with at least one of the following general symptoms: fever or low-grade fever, malaise, headache and myalgia; and at least one of the following three respiratory symptoms: cough, odynophagia and/or dyspnea. The VIGIRA network registers the presence of headache consistently. During the 2021/2022 season, the prevalence rate of influenza-like illness was estimated in 758 per 100,000 inhabitants.

In the VIGIRA program all patients who meet definition criteria are registered as cases (clinical cases). Among these, the sentinels take between 2 and 4 samples of nasopharyngeal swab with a sterile swab. Sampling is done in some patients that consult within 5 days from the beginning of the symptoms, especially if fever is one of the clinical symptoms, to ensure a sufficient viral load. The samples are sent to the reference laboratories, where molecular analysis is performed by polymerase chain reaction (PCR) to detect influenza viruses or other respiratory pathogens. All of those samples with a positive influenza result are sent to the CNG for confirmation, sequencing and cultivation.

Methods:

1. Headache prevalence during the course of the infection:

   1. Data from the VIGIRA program database will be processed and analyzed for the influenza seasons between 2010 and 2022. The proportion of patients who presented headache during each flu season will be estimated.
   2. Data obtained during the 2022-2023 and 2023-2024 flu seasons will be estimated by a systematic evaluation of all consecutive patients with a microbiological confirmation of the infection. A telephone-based evaluation will be carried out on all the incident cases that are notified to the VIGIRA network. All patients will be informed about the study objectives and invited to participate. In these patients who consent to participate, a structured questionnaire will be administered, including questions about whether they experienced headache during the course of the influenza infection.

   In both cases, the 95% confidence interval will be calculated and a stratified analysis will be performed for the secondary and exploratory objectives.
2. Factors associated with the presence of headache:

   The variables available in the VIGIRA system database in the historical series 2010-2022 will be analyzed, including:

   A) Demographic data: age, sex. B) Personal history: diabetes/metabolic disease, smoking, obesity, cardiovascular disease, chronic obstructive pulmonary disease, neoplasia or immunosuppression, chronic kidney disease, chronic liver disease, pregnancy, and vaccination status.

   C) Symptoms experienced during influenza infection: fever, shivers, asthenia, myalgia, pain in a localization other than headache, cough, dyspnea, nasal erythema, pharyngeal mucosa erythema, headache, or gastrointestinal symptoms. Also, other features, such as sudden onset of the symptoms, and the exposure to another person infected with influenza will be assessed.

   D) Variables related to the disease course and prognosis: these will include the need of referral to a specialized center; the presence of otitis, sinusitis, pneumonia; and all-cause death. The specific influenza strain will be described, as well.

   A logistic regression analysis will be performed in which the dependent variable will be the presence of headache. Those variables that in the univariate analysis present a P value lower than 0.1 will be included in a Multivariate analysis. Compensation for multiple comparisons will be made through the procedure of False Discovery Rate with the process of Benjamini-Hochberg, and those variables with a P value lower than 0.05 will be considered statistically significant.
3. Differences in the prognosis depending on the presence of headache:

   The variables available in the VIGIRA base from the historical series from 2010-2022 listed in the section 2 will be used.

   Three logistic regression analyses will be performed, in which the dependent variables will be death, need of hospitalization and presence of pneumonia. A reproduction of the model performed and detailed in the point 2 will be made. In all three cases, it will be evaluated whether the presence of headache, after adjusting for those variables that may act as confounding factors, is associated with a different prognosis. Those parameters listed in the exploratory objectives will also be evaluated.
4. Clinical characterization of the headache phenotype of headache attributed to Influenza infection:

   During the 2022-2023 flu season, a prospective cohort study will be conducted. All consecutive cases with a microbiological diagnosis of influenza infection will be contacted by a trained evaluator, who will collect the data directly in an anonymized database. An evaluator will contact the patients within 14 days after the start of the symptoms, with the aim of: 1) Having sufficient time of evolution of the disease to evaluate its clinical expressiveness and the duration of the headache; 2) Allow the responsible primary care physician to communicate the diagnosis to the patient and the therapeutic measures to be adopted; 3) Minimize the memory bias that would imply a more delayed evaluation.

   The following variables will be included:

   A) Demographic data: Age in the moment of the infection, sex, ethnicity.

   B) Prior medical history: Hypertension, diabetes, smoking, cardiological disorders, respiratory, immunological, oncological, or neurological disorders. Prior history of primary headache and prior episodes of headache in the context of other infections will be assessed, including the source of the diagnosis (general practitioner, neurologist, other), and a positive family history of headache. The vaccination status to prevent influenza will be assessed, including the vaccination date and the specific vaccine.

   C) Headache-related data: days elapsed between the symptom onset and the headache onset, duration of headache, circadian pattern of the headache, association between the headache and the presence of fever, location of headache (holocranial, hemicranial), topography (frontal, temporal, parietal, occipital, vertex, facial, cervical and/or periocular), pain quality (presence of oppressive, stabbing, throbbing, burning, electric or others), headache intensity (verbal analog scale 0-10, 0: no pain, 10: worst possible pain), presence of other symptoms (photophobia, phonophobia, osmophobia, nausea, vomiting, worsening by physical activity, avoidance of physical activity, cranial autonomic symptoms), presence of other neurological symptoms (blurred vision, tingling, loss of strength or altered sensorium), association of the headache with postural changes, disability generated by the headache (proportion of daily activities that could not be performed on a 0-100 scale, being 0 none and 100 all). The presence of red flags will be systematically assessed, including wake-up headache, progressive worsening, resistance to symptomatic treatment, judgment as the worst headache ever experienced, sudden onset of the headache, confusion, and decreased level of consciousness). The need, modality and outcome of acute treatment will be evaluated.

   D) Symptoms experienced during the infection: The following symptoms will be systematically assessed: anosmia, arthralgia, asthenia, weakness, diarrhea, dyspnea, pain thoracic, expectoration, fever, dizziness, myalgia, odynophagia, rash, runny nose, cough, vomiting, syncope, dysgeusia.

   E) Variables related to the prognosis (presence of pneumonia, need for oxygen therapy, admission to the intensive care unit).

   A comparison will be made between the mentioned variables in the subgroups included in the exploratory objectives: sex, vaccination status, circulating influenza strain, and presence of microbiological confirmation.
5. Duration of the headache in patients that suffer from it as a symptom of the influenza infection.

In these patients in which the headache persists by the time of the clinical evaluation, a prospective follow-up will be done. Patients will be contacted by phone every other week until the headache resolution. A description of headache duration using the Kaplan-Meier survival method will be done. The following subgroups will be assessed: female sex, state of vaccination, and circulating strain.

To evaluate which variables are associated to a longer duration of the headache, a cox-regression analysis will be carried out. First, a univariate analysis will be conducted, and those variables that are associated with a different duration of the headache and present a P-value lower than 0.2 t will be included in a multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of influenza virus infection, using molecular techniques (PCR) or antigen test.
2. Age older than 18 years old.

Exclusion Criteria:

1. Critical medical situation that makes impossible the clinical interview and evaluation of clinical symptoms.
2. Prior history of dementia or cognitive impairment that makes it difficult to assess patients or describe symptoms.
3. Speech or language impairment, or insufficient comprehension of the Spanish language that makes evaluation difficult.
4. Deceased during the course of the flu infection before they could be tested.
5. Decline to be interviewed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with a confirmed influenza infection. Patients belonging to a general practitioner or sentinel pediatrician quota who are evaluated in primary care (PC) by an IRA. Sample collection is performed in some patients who consult within 5 days from the onset of symptoms, especially if there is a clinical picture of fever.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of headache as an influenza symptom | During each influenza season, starting on the season 2010 and until the season 2022, an average of 1 year per season
  To calculate the proportion of patients who reported headache during the course of influenza infection

SECONDARY OUTCOMES:
Prevalence of headache as an influenza symptom - prospective | During the 2022-2024 influenza seasons, an average of 1 year per season
  Prospective evaluation of prevalence of headache, after interviewing all consecutive patients, during the 2022-2024 influenza seasons
Predictors of headache as an influenza symptom | Including data from influenza seasons 2010-2022, an average of 1 year per season
  Demographic or clinical variables are associated with the presence of headache in patients with influenza infection in a logistic regression analysis (dependent variable: headache)
Predictors of headache as an influenza symptom - prospective | During the 2022-2024 influenza seasons, an average of 1 year per season
  Demographic or clinical variables are associated with the presence of headache in patients with influenza infection in a logistic regression analysis (dependent variable: headache)
Impact of headache in the prognosis of influenza | Including data from influenza seasons 2010-2022, an average of 1 year per season
  Three logistic regression analyses will be performed, in which the dependent variables will be death, need of hospitalization and presence of pneumonia. In all three cases, it will be evaluated whether the presence of headache, after adjusting for those variables that may act as confounding factors, is associated with a different prognosis
Impact of headache in the prognosis of influenza - prospective | During the 2022-2024 influenza seasons, an average of 1 year per season
  Three logistic regression analyses will be performed, in which the dependent variables will be death, need of hospitalization and presence of pneumonia. In all three cases, it will be evaluated whether the presence of headache, after adjusting for those variables that may act as confounding factors, is associated with a different prognosis
Clinical phenotype of headache during the course of influenza | During the influenza seasons 2022-2024, an average of 1 year per season
  To characterize the headache phenotype and the presence of specific and distinctive features and its differentiation from other headache disorders based on the presence of red flags
Prospective evaluation of the duration of headache during the course of influenza | During the influenza seasons 2022-2024, an average of 1 year per season
  Patients with persistent headache by the time of the clinical interview will be prospectively followed up. Patients will be contacted by phone every other week until the headache resolution

OTHER OUTCOMES:
Sex-adjusted prevalence of headache as an influenza symptom | During the influenza seasons 2010-2022, an average of 1 year per season
  To compare the proportion of patients who report headache during the course of influenza infection between female and male patients
Sex-adjusted prevalence of headache as an influenza symptom - prospective | During the influenza seasons 2022-2024, an average of 1 year per season
  To compare the proportion of patients who report headache during the course of influenza infection between female and male patients.
Age-adjusted prevalence of headache as an influenza symptom | During the influenza seasons 2010-2022, an average of 1 year per season
  To compare the proportion of patients who report headache during the course of influenza infection within the different age groups.
Age-adjusted prevalence of headache as an influenza symptom - prospective | During the influenza seasons 2022-2024, an average of 1 year per season
  To compare the proportion of patients who report headache during the course of influenza infection within the different age groups.
Vaccination-adjusted prevalence of headache as an influenza symptom | During the influenza seasons 2010-2022, an average of 1 year per season
  To compare the proportion of patients who report headache during the course of influenza infection depending on the vaccination status of patients
Vaccination-adjusted prevalence of headache as an influenza symptom - prospective | During the influenza seasons 2022-2024, an average of 1 year per season
  To compare the proportion of patients who report headache during the course of influenza infection depending on the vaccination status of patients.
Influenza strain-adjusted prevalence of headache as an influenza symptom | During the influenza seasons 2010-2022, an average of 1 year per season
  To compare the proportion of patients who report headache during the course of influenza infection depending on the circulating influenza strain(s) of each season.
Influenza strain-adjusted prevalence of headache as an influenza symptom - prospective | During the influenza seasons 2022-2024, an average of 1 year per season
  To compare the proportion of patients who report headache during the course of influenza infection depending on the circulating influenza strain(s) of each season.

CONTACTS AND LOCATIONS:
Overall Officials: David García Azorín, MD, PhD, Principal Investigator — Sanidad de Castilla y León
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared upon reasonable request to the principal investigator.

REFERENCES:
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Fendrick AM, Monto AS, Nightengale B, Sarnes M. The economic burden of non-influenza-related viral respiratory tract infection in the United States. Arch Intern Med. 2003 Feb 24;163(4):487-94. doi: 10.1001/archinte.163.4.487. PMID 12588210
- [Background] Iuliano AD, Roguski KM, Chang HH, Muscatello DJ, Palekar R, Tempia S, Cohen C, Gran JM, Schanzer D, Cowling BJ, Wu P, Kyncl J, Ang LW, Park M, Redlberger-Fritz M, Yu H, Espenhain L, Krishnan A, Emukule G, van Asten L, Pereira da Silva S, Aungkulanon S, Buchholz U, Widdowson MA, Bresee JS; Global Seasonal Influenza-associated Mortality Collaborator Network. Estimates of global seasonal influenza-associated respiratory mortality: a modelling study. Lancet. 2018 Mar 31;391(10127):1285-1300. doi: 10.1016/S0140-6736(17)33293-2. Epub 2017 Dec 14. PMID 29248255
- [Background] Perez-Rubio A, Platero L, Eiros Bouza JM. Seasonal influenza in Spain: Clinical and economic burden and vaccination programmes. Med Clin (Barc). 2019 Jul 5;153(1):16-27. doi: 10.1016/j.medcli.2018.11.014. Epub 2019 Jan 6. English, Spanish. PMID 30621906
- [Background] Redondo-Bravo L, Delgado-Sanz C, Oliva J, Vega T, Lozano J, Larrauri A; Spanish Influenza Sentinel Surveillance System. Transmissibility of influenza during the 21st-century epidemics, Spain, influenza seasons 2001/02 to 2017/18. Euro Surveill. 2020 May;25(21):1900364. doi: 10.2807/1560-7917.ES.2020.25.21.1900364. PMID 32489178
- [Background] Ortiz de Lejarazu Leonardo R, Rojo Rello S, Sanz Munoz I. Diagnostic challenges in influenza. Enferm Infecc Microbiol Clin (Engl Ed). 2019 May;37 Suppl 1:47-55. doi: 10.1016/S0213-005X(19)30182-X. English, Spanish. PMID 31138423
- [Background] Brody H. Influenza. Nature. 2019 Sep;573(7774):S49. doi: 10.1038/d41586-019-02750-x. No abstract available. PMID 31534258
- [Background] Eccles R. Mechanisms of symptoms of the common cold and influenza. Br J Hosp Med (Lond). 2007 Feb;68(2):71-5. doi: 10.12968/hmed.2007.68.2.22824. No abstract available. PMID 17370703
- [Background] Eccles R. Understanding the symptoms of the common cold and influenza. Lancet Infect Dis. 2005 Nov;5(11):718-25. doi: 10.1016/S1473-3099(05)70270-X. PMID 16253889
- [Background] Pedersen CJ, Quinn JV, Rogan DT, Yang S. Factors Associated With Influenza in an Emergency Department Setting. J Emerg Med. 2019 May;56(5):478-483. doi: 10.1016/j.jemermed.2018.12.012. Epub 2019 Feb 22. PMID 30803847
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Trigo J, Garcia-Azorin D, Planchuelo-Gomez A, Martinez-Pias E, Talavera B, Hernandez-Perez I, Valle-Penacoba G, Simon-Campo P, de Lera M, Chavarria-Miranda A, Lopez-Sanz C, Gutierrez-Sanchez M, Martinez-Velasco E, Pedraza M, Sierra A, Gomez-Vicente B, Arenillas JF, Guerrero AL. Factors associated with the presence of headache in hospitalized COVID-19 patients and impact on prognosis: a retrospective cohort study. J Headache Pain. 2020 Jul 29;21(1):94. doi: 10.1186/s10194-020-01165-8. PMID 32727345
- [Background] Garcia-Azorin D, Sierra A, Trigo J, Alberdi A, Blanco M, Calcerrada I, Cornejo A, Cubero M, Gil A, Garcia-Iglesias C, Lozano AG, Martinez Badillo C, Montilla C, Mora M, Nunez G, Paniagua M, Perez C, Rojas M, Ruiz M, Sierra L, Hurtado ML, Guerrero Peral AL. Frequency and phenotype of headache in covid-19: a study of 2194 patients. Sci Rep. 2021 Jul 19;11(1):14674. doi: 10.1038/s41598-021-94220-6. PMID 34282206
- [Background] Caronna E, Ballve A, Llaurado A, Gallardo VJ, Ariton DM, Lallana S, Lopez Maza S, Olive Gadea M, Quibus L, Restrepo JL, Rodrigo-Gisbert M, Vilaseca A, Hernandez Gonzalez M, Martinez Gallo M, Alpuente A, Torres-Ferrus M, Pujol Borrell R, Alvarez-Sabin J, Pozo-Rosich P. Headache: A striking prodromal and persistent symptom, predictive of COVID-19 clinical evolution. Cephalalgia. 2020 Nov;40(13):1410-1421. doi: 10.1177/0333102420965157. PMID 33146036
- [Background] Gonzalez-Martinez A, Fanjul V, Ramos C, Serrano Ballesteros J, Bustamante M, Villa Marti A, Alvarez C, Garcia Del Alamo Y, Vivancos J, Gago-Veiga AB. Headache during SARS-CoV-2 infection as an early symptom associated with a more benign course of disease: a case-control study. Eur J Neurol. 2021 Oct;28(10):3426-3436. doi: 10.1111/ene.14718. Epub 2021 Feb 2. PMID 33417287
- [Background] Trigo J, Garcia-Azorin D, Sierra-Mencia A, Tamayo-Velasco A, Martinez-Paz P, Tamayo E, Guerrero AL, Gonzalo-Benito H. Cytokine and interleukin profile in patients with headache and COVID-19: A pilot, CASE-control, study on 104 patients. J Headache Pain. 2021 Jun 4;22(1):51. doi: 10.1186/s10194-021-01268-w. PMID 34088273
- [Background] Lopez JT, Garcia-Azorin D, Planchuelo-Gomez A, Garcia-Iglesias C, Duenas-Gutierrez C, Guerrero AL. Phenotypic characterization of acute headache attributed to SARS-CoV-2: An ICHD-3 validation study on 106 hospitalized patients. Cephalalgia. 2020 Nov;40(13):1432-1442. doi: 10.1177/0333102420965146. PMID 33146037
- [Background] Garcia-Azorin D, Trigo J, Talavera B, Martinez-Pias E, Sierra A, Porta-Etessam J, Arenillas JF, Guerrero AL. Frequency and Type of Red Flags in Patients With Covid-19 and Headache: A Series of 104 Hospitalized Patients. Headache. 2020 Sep;60(8):1664-1672. doi: 10.1111/head.13927. Epub 2020 Aug 18. PMID 32790215
- [Background] Planchuelo-Gomez A, Trigo J, de Luis-Garcia R, Guerrero AL, Porta-Etessam J, Garcia-Azorin D. Deep Phenotyping of Headache in Hospitalized COVID-19 Patients via Principal Component Analysis. Front Neurol. 2020 Dec 17;11:583870. doi: 10.3389/fneur.2020.583870. eCollection 2020. PMID 33391152
- [Background] Garcia-Azorin D, Layos-Romero A, Porta-Etessam J, Membrilla JA, Caronna E, Gonzalez-Martinez A, Mencia AS, Segura T, Gonzalez-Garcia N, Diaz-de-Teran J, Gallardo VJ, Gago-Veiga AB, Ballve A, Trigo Lopez J, Sastre-Real M, Llaurado A, Cornejo A, de Lorenzo I, Guerrero-Peral A, Pozo-Rosich P. Post-COVID-19 persistent headache: A multicentric 9-months follow-up study of 905 patients. Cephalalgia. 2022 Jul;42(8):804-809. doi: 10.1177/03331024211068074. Epub 2022 Feb 15. PMID 35166156
- [Derived] Garcia-Azorin D, Santana-Lopez L, Lozano-Alonso JE, Ordax-Diez A, Gonzalez-Osorio Y, Rojo-Rello S, Eiros JM, Sanchez-Martinez J, Recio-Garcia A, Sierra-Mencia A, Sanz-Munoz I, Guerrero-Peral AL. InfluenCEF study: Clinical phenotype and duration of headache attributed to influenza infection. Cephalalgia. 2023 Nov;43(11):3331024231212900. doi: 10.1177/03331024231212900. PMID 37950674
- See also: Boletín informativo de la Red Centinela Sanitaria de Castilla y León, 2022 — https://www.saludcastillayleon.es/profesionales/es/centinelas/informes-boletines-red-centinela-sanitaria-castilla-leon.ficheros/2159835-Bolet%C3%ADn%202022%20n%C2%BA%201.pdf
- See also: World Health Organization Europe. WHO Regional Office for Europe guidance for sentinel influenza surveillance inhumans. May 2011. — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&ved=2ahUKEwjPyY3Tvo_8AhWyg_0HHdFDAeYQFnoECBUQAQ&url=https%3A%2F%2Fwww.euro.who.int%2F__data%2Fassets%2Fpdf_file%2F0020%2F90443%2FE92738.pdf&usg=AOvVaw2XfAlgGn9lDjXZ61T5EeZH